CLINICAL TRIAL: NCT04667845
Title: Digital Home Ovulation Test One Cycle at Home Study
Status: Completed | Type: Observational
Sponsor: SPD Development Company Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PROTOCOL-1200
Record Dates: First submitted 2020-12-08; First posted 2020-12-16 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Pregnancy; Fertility
Keywords: Trying to Conceive; Digital Home Ovulation Test; Usability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Home Ovulation Test — Digital read home ovulation test

SUMMARY:
This study will assess the usability of a Digital Home Ovulation Test when used at home by lay-users seeking to conceive.

DETAILED DESCRIPTION:
This study will assess the ease of use of a Digital Home Ovulation Test when used by lay-users for one cycle in their home environment. The home ovulation test to be used in the study is a digital home ovulation test used to detect luteinising hormone (LH) and Estrone-3-Glucuronide (E3G) in urine to identify when ovulation is imminent.

A sample size of 120 volunteers (minimum) will provide adequate information for assessing the usability of the home ovulation test. Usability of the test will be assessed through a questionnaire completed at the end of the study.

This observational study will be conducted remotely and volunteers representative of the intended user (lay-users) will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18 to 45 years
* Seeking to conceive
* Willing to give informed consent and comply with the investigational procedures

Exclusion Criteria:

* Taking medication, or has known condition which means they should not get pregnant.
* Currently pregnant or breastfeeding
* Used the digital ovulation test within the last six months
* Currently or previously employed by Swiss Precision Diagnostics (SPD), Abbott, Alere, Unipath, P&G or affiliates
* Has an immediate* relative currently or previously (within past 5 years) employed by SPD, Abbott, Alere, Unipath or P&G, or affiliates

  *Immediate relatives are defined as parents, children, siblings or partner/spouse
* Is a qualified or trainee healthcare professional (HCP)
* Has professional experience of using dipstick type tests or lateral flow devices
* Using any treatment which may affect the menstrual cycle (e.g. contraceptive pill)
* Using infertility medications or hormone replacement medications containing Luteinising Hormone (LH) or Human Chorionic Gonadotrophin (hCG) (e.g. Pregnyl®)
* Using or undergoing any other medical treatment for fertility such as ovulation drugs, artificial insemination and assisted fertility such as In vitro fertilization (IVF) or Intracytoplasmic sperm injection (ICSI)
* Peri-or post-menopausal, e.g. experiencing symptoms: irregular menstrual periods, hot flushes, night sweats, sleep disturbances and/or moods swings
* Has been diagnosed with polycystic ovarian syndrome (PCOS)
* Has PCOS symptoms e.g. very irregular cycles, hirsutism
* Has abnormal liver or kidney function
* Is taking antibiotics containing tetracycline

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women seeking to conceive
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2021-04-22 (Actual)

PRIMARY OUTCOMES:
Device usability | One menstrual cycle, average 28 days
  The usability of the digital home ovulation test when used at home by volunteers seeking to conceive scored on a 7 point Likert scale where 1 is the lowest (most negative) score and 7 is the highest (most positive) score.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Johnson, Study Director — SPD Development Company
Locations (1):
- SPD Development Company Ltd, Bedford, Bedfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No